CLINICAL TRIAL: NCT01285921
Title: Functional Link Between Hippocampal and Vestibular Systems: a Pilot Study in Epilepsy Surgery Principal Investigator: Elizabeth VITTE
Brief Title: Functional Link Between Hippocampal and Vestibular Systems: a Pilot Study in Epilepsy Surgery
Acronym: HIPPOCAMPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: P100106; 2010-A01220-39 (Other: IDRCB)
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
Keywords: hippocampal; vestibular test
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- hippocampal surgery (Experimental): Vestibular test before and after hippocampal surgery
  Principal criterion:
  Research for an asymmetry of the vestibular responses (Caloric test, Vestibular Evoked Myogenic potentials: VEMp, Head Impulse Test: HIT, Eye Rotational Test: ERI). Investigator performs a blind vestibular test (single blind)
  Interventions: Other: vestibular test before and after hippocampal surgery

INTERVENTIONS:
Other: vestibular test before and after hippocampal surgery — * Research of a spontaneous nystagmus with and without fixation(VIDEONYSTAGMOSCOPY) and segmentary deviations (Fukuda test)
  * HIT (testing semicircular canal function at high frequency).Results: Gain in %
  * VEMp (testing saccular function). Results: Amplitude in μV and latency in ms
  * ERI (testing lateral semicircular function at middle frequency). Results: Nystagmus during and after the rotations in frequency and slow phase velocity (SPV) in °/s
  * Caloric test (testing lateral semicircular function at low frequency). Results: Canal paresis in % and SPV in °/S

SUMMARY:
Vestibular signals deeply influence hippocampal spatial representations and may contribute to the navigational deficits of humans with vestibular dysfunction. The reciprocal influence of hippocampal signals on the vestibular system are more putative. The investigators wish to investigate in this pilot study the consequences on vestibular system of the removal of the hippocampal formation to treat drug resistant temporal lobe epilepsy.

DETAILED DESCRIPTION:
Functional link between hippocampal and vestibular systems: a pilot study in epilepsy surgery

Hypothesis:

The human hippocampal formation plays a crucial role in various aspects of memory processing. Work in rodents and some other species emphasized the role of the hippocampus in spatial learning and memory as well. A few human studies also point to a direct relation between hippocampal size, navigation and spatial memory. Patients with acquired chronic bilateral vestibular loss develop a significant selective atrophy of the hippocampus (Brandt et al, 2005) and activation of lateral semicircular canal by caloric stimulation induces activation of hippocampal formation in f-MRI (VITTE et al, 1996). But the investigators still do not know the effects on vestibular responses of the removal of the hippocampal formation to cure temporal lobe epilepsy. If the hippocampal formation directly influences the vestibular response, an asymmetry of the vestibular responses should be recorded postoperatively.

Principal criterion Research for an asymmetry of the vestibular responses (Caloric test, Vestibular Evoked Myogenic potentials: VEMp, Head Impulse Test: HIT, Eye Rotational Test: ERI)

Inclusion criteria

* patients suffering of intractable mesial temporal lobe epilepsy and candidate for surgery,
* without history of any cochlea-vestibular disorder
* older than 18 years,
* French residents,
* with medicare,
* after signed informed consent. Exclusion criteria
* History of cochlea-vestibular disorder
* Pregnancy

Population

* 22 patients suffering of intractable epilepsy and candidate for surgery (10 right side and 10 left side).
* Evaluation before and after surgery

Methodology Vestibular function will be quantified by daily practice vestibular tests

* Research of a spontaneous nystagmus with and without fixation (VIDEONYSTAGMOSCOPY) and segmentary deviations (Fukuda test)
* HIT (testing semicircular canal function at high frequency). Results: Gain in %
* VEMp (testing saccular function). Results: Amplitude in μV and latency in ms
* ERI (testing lateral semicircular function at middle frequency). Results: Nystagmus during and after the rotations in frequency and slow phase velocity (SPV) in °/s
* Caloric test (testing lateral semicircular function at low frequency). Results: Canal paresis in % and SPV in °/S

Results Vestibular function will be quantified with daily practice vestibular tests

* Quantification of the vestibular asymmetry
* Ipsi or contralateral to the side of the surgery?
* Depending on the hemispheric dominance?

ELIGIBILITY:
Inclusion Criteria:

* patients suffering of intractable mesial temporal lobe epilepsy and candidate for surgery,
* without history of any cochlea-vestibular disorder
* older than 18 years,
* French residents,
* with medicare,
* after signed informed consent

Exclusion Criteria:

* History of cochlea-vestibular disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
caloric test | 6 months after surgery
  -Caloric test (testing lateral semicircular function at low frequency). Results: Canal paresis in % and SPV in °/S

SECONDARY OUTCOMES:
vestibular test | 6 months after surgery
  * Research of a spontaneous nystagmus with and without fixation(videonystagmoscopy) and segmentary deviations (Fukuda test)
  * HIT (testing semicircular canal function at high frequency). Results: Gain in %
  * VEMp (testing saccular function). Results: Amplitude in μV and latency in ms
  * ERI (testing lateral semicircular function at middle frequency). Results: Nystagmus during and after the rotations in frequency and slow phase velocity (SPV) in °/s

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Vitte, MD, PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital BEAUJON, Clichy, France

IPD SHARING:
Plan to Share IPD: No